CLINICAL TRIAL: NCT07060248
Title: A Study Based on CT Radiomics for Distinguishing Benign From Malignant Renal Tumors and Assessing Their Aggressiveness.
Status: Active, not recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: JLiu
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RCC group, non-RCC group; WHO/ISUP low-grade ccRCC, high-grade ccRCC; T3 tumor, T1-T2 tumor

SUMMARY:
To evaluate the efficacy of CT-based radiomics in differentiating benign from malignant renal tumors, predicting nuclear grading of renal cell carcinoma, and assessing T-stage of renal tumors, thereby exploring its clinical application value.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed renal tumors (including clear cell renal cell carcinoma, papillary renal cell carcinoma, chromophobe renal cell carcinoma, angiomyolipoma, and oncocytoma).
* Contrast-enhanced CT scan was performed preoperatively.

Exclusion Criteria:

* Pure cystic clear cell renal cell carcinoma
* Poor-quality CT images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal mass
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
CT-based radiomics analysis for benign and malignant tumor differentiation | within 1 month
  Histopathological diagnosis served as the gold standard, with tumors classified into: (1) Benign renal tumors: Including lipid-poor angiomyolipoma and renal oncocytoma; (2) Malignant renal tumors: Comprising clear cell renal cell carcinoma, papillary renal cell carcinoma, and chromophobe renal cell carcinoma
CT-based radiomics analysis for nuclear grading of clear cell renal cell carcinoma (ccRCC) | within 1 month
  Histopathological diagnosis served as the gold standard, with tumors classified into: (1) low grade ccRCC: Including WHO/ISUP grade 1-2 ccRCC; (2) high grade ccRCC: Including WHO/ISUP grade 3-4 ccRCC
CT-based radiomics analysis of T-stage classification of renal cell carcinoma (RCC) | within 1 month
  Histopathological diagnosis served as the gold standard, with tumors classified into: (1) low T-stage RCC: Including T1-2 RCC; (2) high T-stage RCC: including T3-4 RCC

CONTACTS AND LOCATIONS:
Locations (1):
- Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The original data were not publicly available and could only be shared with the permission of the local ethics committee.